CLINICAL TRIAL: NCT06157424
Title: Evaluating Efficacy and Safety of Combined Thread Embedding and Auricular Acupuncture in Gastroesophageal Reflux Disease With Liver Qi Invading Stomach Pattern: A Randomized Controlled Trial
Brief Title: Efficacy and Safety of Combined Thread Embedding Acupuncture With Auricular Acupuncture for GERD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Bui Pham Minh Man, Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 703/HDDD-DHYD
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture + Standard treatment (Experimental): Standard treatment plus thread embedding acupuncture and auricular acupuncture
  Interventions: Other: Thread Embedding Acupuncture; Other: Auricular acupuncture; Other: Standard treatment
- Standard treatment (Active Comparator): Standard treatment
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Thread Embedding Acupuncture — Thread Embedding Acupuncture is applied at acupoints including CV-12, CV-13, ST-36, PC-6, BL-17, BL-18, BL-21 on both sides of the body every 2 weeks, totaling 2 sessions over 4 weeks of intervention.
  Arms: Acupuncture + Standard treatment
Other: Auricular acupuncture — Auricular acupuncture is administered using adhesive patches with small needles (0.25 x 1.3 mm) placed at acupoints TF4, AH6, CO12, CO4, CO2 once a week, totaling 4 sessions over the 4-week intervention period.
  Arms: Acupuncture + Standard treatment
Other: Standard treatment — Standard treatment, continuously administered over the 4-week intervention period, involves standard doses of proton pump inhibitors, additional antacids as needed, and lifestyle modifications.

SUMMARY:
Gastroesophageal reflux disease (GERD) is increasingly prevalent today. Proton-pump inhibitors (PPIs) are the primary treatment, yet their effectiveness remains limited. Various acupuncture methods have shown promise in treating GERD. Among these, thread embedding acupuncture (TEA) and auricular acupuncture (AA) offer the advantage of prolonged treatment per intervention, significantly reducing healthcare visits for procedures, particularly beneficial for conditions requiring extended therapy. This has led to the widespread application of TEA and AA in GERD treatment. However, evidence supporting their effectiveness remains inconclusive. In this study, we aim to assess the efficacy and safety of combining TEA with AA for treating GERD. According to traditional medicine, treatment should be pattern-based. Thus, we will focus on patients exhibiting the Liver Qi Invading Stomach pattern, as reports indicate its prevalence among GERD patients.

DETAILED DESCRIPTION:
Patients with GERD diagnosed through the GerdQ score and presenting the traditional medicine pattern of Liver Qi invading Stomach, meeting the inclusion and not the exclusion criteria, will be included in the study. Upon randomization, participants will be allocated into two groups: the control and intervention groups.

The study spans four weeks. Both groups will receive standard GERD treatment following current guidelines, which include PPIs, additional antacids as required, and lifestyle modifications. The intervention group will receive an additional combination of thread embedding acupuncture therapy (TEA) every other week and auricular acupuncture (AA) weekly.

Patients will undergo weekly follow-up examinations. Symptom assessment, quality of life evaluations using specific questionnaires, and antacid medication usage will be monitored weekly. Adverse effects (AE) related to the treatment will be documented throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged from 18 to 60 Years
* GerdQ score of eight or higher
* Having heartburn and/or regurgitation on two days per week or more
* Diagnosis of GERD with Liver Qi Invading Stomach Pattern

Exclusion Criteria:

* Any prior endoscopy-confirmed structural diseases
* Uncontrolled inflammatory bowel disease, chronic or genetic conditions, alcohol or drug abuse history
* Alarming symptoms indicating gastric cancer, complicated ulcers, or serious illnesses
* History of esophageal or gastrointestinal surgery
* Current use of medications impacting GERD treatment or assessment
* Recent (within two weeks) Western Medicine or Traditional Medicine treatment for GERD
* History of hypersensitivity reactions to any components involved in the intervention
* Pregnancy or breastfeeding
* Current participation in any other clinical trials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
The proportion of heartburn resolution | Day 0 and after every week during 4-week treatment (day 0, day 7, day 14, day 21, day 28)
  Heartburn resolution is assessed through patient inquiry during each follow-up examination.

SECONDARY OUTCOMES:
The proportion of regurgitation resolution | Day 0 and after every week during 4-week treatment (day 0, day 7, day 14, day 21, day 28)
  Regurgitation resolution is assessed through patient inquiry during each follow-up examination.
Chang in the Gastroesophageal Reflux disease Questionnaire (GerdQ) score | Day 0 and after every week during 4-week treatment (day 0, day 7, day 14, day 21, day 28)
  As per GerdQ, patients were prompted to recall their symptoms and utilization of over-the-counter medications in the past week. It employs a four-point Likert scale (0-3) for scoring, resulting in a total GerdQ score range from 0 to 18. A higher score signifies a more severe condition.
Chang in the Frequency Scale for the Symptoms of GERD (FSSG) score | Day 0 and after every two week during 4-week treatment (day 0, day 14, day 28)
  The FSSG questionnaire consists of twelve questions categorized into two domains: reflux symptoms and dysmotility symptoms. Using a 5-point Likert scale (0-4), the FSSG yields a total score range of 0 to 48. A higher score suggests a more severe or significant disease.
Chang in the Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) score | Day 0 and after every two week during 4-week treatment (day 0, day 14, day 28)
  The GERD-HRQL questionnaire consists of 16 questions utilizing a numerical Likert-type response. Patients assess symptom severity on an ordinal scale ranging from 0 to 5. The total score range for GERD-HRQL spans from 0 to 80, incorporating evaluations for heartburn, regurgitation, and other related aspects. A higher score reflects a more severe disease.
Changes in the number of antacid packets used | Day 0 and after every week during 4-week treatment (day 0, day 7, day 14, day 21, day 28)
  The number of antacid packets used per week will be recorded during each follow-up visit.
The proportion of side effects of thread embedding acupuncture and auricular acupuncture | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medical Center HCMC - Branch no.3, University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Maret-Ouda J, Markar SR, Lagergren J. Gastroesophageal Reflux Disease: A Review. JAMA. 2020 Dec 22;324(24):2536-2547. doi: 10.1001/jama.2020.21360. PMID 33351048
- [Background] Luo Z, Hu X, Chen C, Zhu L, Zhang W, Shen Y, He J. Effect of Catgut Embedment in Du Meridian Acupoint on Mental and Psychological Conditions of Patients with Gastroesophageal Reflux Disease. Evid Based Complement Alternat Med. 2020 Sep 22;2020:5415813. doi: 10.1155/2020/5415813. eCollection 2020. PMID 33029166
- [Background] Katz PO, Gerson LB, Vela MF. Guidelines for the diagnosis and management of gastroesophageal reflux disease. Am J Gastroenterol. 2013 Mar;108(3):308-28; quiz 329. doi: 10.1038/ajg.2012.444. Epub 2013 Feb 19. No abstract available. PMID 23419381
- [Background] Hunt R, Armstrong D, Katelaris P, Afihene M, Bane A, Bhatia S, Chen MH, Choi MG, Melo AC, Fock KM, Ford A, Hongo M, Khan A, Lazebnik L, Lindberg G, Lizarzabal M, Myint T, Moraes-Filho JP, Salis G, Lin JT, Vaidya R, Abdo A, LeMair A; Review Team:. World Gastroenterology Organisation Global Guidelines: GERD Global Perspective on Gastroesophageal Reflux Disease. J Clin Gastroenterol. 2017 Jul;51(6):467-478. doi: 10.1097/MCG.0000000000000854. No abstract available. PMID 28591069
- [Background] Sun QH, Li TT, Huang MT, Wang MY, Xiao X, Bai XH. [Acupoint selection rules in treating gastroesophageal reflux disease with acupuncture in China based on data mining]. Zhongguo Zhen Jiu. 2020 Dec 12;40(12):1374-8. doi: 10.13703/j.0255-2930.20191107-0003. Chinese. PMID 33415885
- [Background] Zhu J, Guo Y, Liu S, Su X, Li Y, Yang Y, Hou L, Wang G, Zhang J, Chen JJ, Wang Q, Wei R, Wei W. Acupuncture for the treatment of gastro-oesophageal reflux disease: a systematic review and meta-analysis. Acupunct Med. 2017 Oct;35(5):316-323. doi: 10.1136/acupmed-2016-011205. Epub 2017 Jul 8. PMID 28689187
- [Background] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213